CLINICAL TRIAL: NCT04089839
Title: Prospective Assessment of Dasatinib Management Among CP-CML Patients With Dasatinib Initiation in a Real Life Setting: DasaREALISE.
Brief Title: A Study of Dasatinib Management Among CP-CML (Chronic Phase, Chronic Myeloid Leukemia) Participants Initiating Dasatinib in a Real Life Setting
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-616
Record Dates: First submitted 2019-01-08; First posted 2019-09-13 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CP-CML participants initiating dasatinib
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This is a prospective, non-interventional study conducted in CP-CML patients receiving dasatinib who are enrolled by a sample of hematologists in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than or equal to 18 years
* Patients diagnosed with CP-CML
* Patients who started dasatinib within the last month before inclusion, or on the day of inclusion or within the month after inclusion

Exclusion Criteria:

* Patients participating in an ongoing interventional trial
* Patients diagnosed with AP-CML (accelerated phase) or BP-CML (blast phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All French hematologists will be invited to participate to the study, and the study will be conducted by hematologists agreeing to participate. Each participating investigator will need to enroll consecutive CP-CML patients who meet the selection criteria.
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Incidence of CP-CML patients remaining on dasatinib treatment | 24 months

SECONDARY OUTCOMES:
Distribution of median age of CP-CML patients receiving dasatinib | 24 months
Distribution of sex ratio of CP-CML patients receiving dasatinib | 24 months
Distribution of concomitant treatment of CP-CML patients receiving dasatinib | 24 months
Distribution of cardiovascular risk factors of CP-CML patients receiving dasatinib | 24 months
Distribution of body mass index (BMI) of CP-CML patients receiving dasatinib | 24 months
Distribution of comorbidities of CP-CML patients receiving dasatinib | 24 months
Distribution of disease characteristics duration between diagnosis and drug initiation in CP-CML patients receiving dasatinib | 24 months
Distribution disease characteristics of last known molecular response in CP-CML patients receiving dasatinib | 24 months
SOKAL distribution of disease characteristics of CP-CML patients receiving dasatinib | 24 months
Distribution of prior treatment(s) of CP-CML patients receiving dasatinib | 24 months
Incidence of initiating dasatinib due to suboptimal response | 24 months
Incidence of initiating dasatinib due to failure | 24 months
Incidence of initiating dasatinib due to intolerance | 24 months
Incidence of initiating dasatinib due to convenience | 24 months
Incidence of initiating dasatinib due to physician decision | 24 months
Incidence of AE's | 24 months
Incidence of SAE's | 24 months
Utilization of dasatinib | 24 months
Incidence of complete molecular response (CMR) | Up to 24 months
Incidence of major molecular response (MMR) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Paris, France

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm